CLINICAL TRIAL: NCT03018665
Title: A Randomized,Active-controlled,Open-label Clinical Trial to Evaluate the Effect of GLP-1 Receptor Agonist (Exenatide Injection) in Combination With Metformin Therapy Compared to Premixed Insulin (BIAsp30) in Combination With Metformin Therapy on Diabetes Remission in Subjects With Newly Diagnosed Type 2 Diabetes Who Are Overweight or Obese
Brief Title: A Study of the Effect of Glucagon-like Peptide 1(GLP-1) Receptor Agonist in Combination With Metformin Therapy on Diabetes Remission in Subjects With Newly Diagnosed Type 2 Diabetes Who Are Overweight or Obese
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Guixia Wang, Director of Endocrinology Department, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JLUEND001
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

ARMS (2):
- Exenatide and Metformin (Experimental): Exenatide in Combination With Metformin
  Interventions: Drug: Exenatide; Drug: Metformin
- BIAsp30 and Metformin (Active Comparator): BIAsp30 in Combination With Metformin
  Interventions: Drug: BIAsp30; Drug: Metformin

INTERVENTIONS:
Drug: Exenatide — subcutaneous injection，5ug twice a day the first month，10ug twice a day the second and third month
  Arms: Exenatide and Metformin
Drug: BIAsp30 — subcutaneous injection，fit dosage twice a day in three months
  Arms: BIAsp30 and Metformin
Drug: Metformin — oral，0.85g，twice a day in three months

SUMMARY:
The purpose of this study is to determine the effect of GLP-1 receptor agonist on inducing diabetes remission in newly diagnosed type 2 diabetes who are overweight or obese

DETAILED DESCRIPTION:
Most of type 2 diabetes are characterized by being overweight or obese mainly caused by insulin resistance. GLP-1 receptor agonist has been proved to help to lose weight and improve insulin resistance. In this study, we suppose that GLP-1 receptor agonist has the effect of inducing diabetes remission in newly diagnosed type 2 diabetes who are overweight or obese and has its advantages

ELIGIBILITY:
Inclusion Criteria:

* A signed and dated informed consent form obtained from the subject before any study related procedures take place.
* Age ≥18 years to ≤65 years at Visit 1.
* The subject has a new diagnosis of type 2 diabetes without any treatment.
* HbA1c ≥8.0% to ≤14.0% at Visit 1.
* BMI(Body Mass Index)≥24kg/m2 to ≤40kg/m2 at Visit 1.

Exclusion Criteria:

* The subject has a history of type 1 diabetes or a secondary form of diabetes.
* The subject has received an anti-diabetic drug before the screening visit.
* Treatment with systemic steroids 2 months prior to screening
* Treatment with anti-obesity drug 2 months prior to screening or any other treatment at the time of screening(i.e. surgery etc) leading to unstable body weight.
* The subject has a history of acute or chronic pancreatitis
* Any gastrointestinal diseases or surgeries that induce chronic malabsorption
* Cancer and medical history of cancer(except basal cell skin cancer or squamous cell skin cancer).
* The subject has a history of recurrent severe hypoglycaemia.
* Cardiovascular disease,within the last 6months prior to screening,defined as: stroke;decompensated heart failure New York Heart Association(NYHA) class III or IV;Myocardial infarction;unstable angina pectoris;or coronary bypass graft or angioplasty.
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure ≥180 millimetre(mm) mercury(Hg) and/or diastolic blood pressure ≥100 millimetre(mm) mercury(Hg).
* Impaired liver function,defined as alanine aminotransferase(ALT) or aspartate aminotransferase(AST) ≥2.5 times upper limit of normal.
* Impaired renal function,defined as serum-creatinine ≥125umol/l for males and ≥110umol/l for females.
* Females who are pregnant or breast-feeding, males and females of childbearing potential,who do not agree to prevent conception during the study.
* Known or suspected abuse of alcohol,narcotics or illicit drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02; Primary Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Inducing Diabetes Remission | At the end of 12-week treatment
Change of Rate of Maintaining Diabetes Remission | 3,6,12,24,36 months after 12-week treatment
Time of Maintaining Diabetes Remission | up to 36 months after 12-week treatment

SECONDARY OUTCOMES:
Change of Blood Pressure | Baseline and 0,3,6,12,24,36 months after 12-week treatment
Change of Heart Rate | baseline and 0,3,6,12,24,36 months after 12-week treatment
Change of Weight | baseline and 0,3,6,12,24,36 months after 12-week treatment
Change of Waistline | baseline and 0,3,6,12,24,36 months after 12-week treatment
Change of Glycosylated Hemoglobin | baseline and 0,3,6,12,24,36 months after 12-week treatment
Change of Pancreatic Beta-cell Function | baseline and 0,3,6,12,24,36 months after 12-week treatment
  Pancreatic Beta-cell Function will be evaluated by insulin releasing test. The fasting and 2-hour postprandial plasma glucose concentrations and serum insulin concentrations will be tested.
Change of Insulin Resistance Index | baseline and 0,3,6,12,24,36 months after 12-week treatment
The Incidence of Hypoglycemia | During the 12-week treatment
The Incidence of Diabetic Retinopathy | up to 36 months after 12-week treatment
The Incidence of Diabetic Nephropathy | up to 36 months after 12-week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guixia Wang, PhD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China